CLINICAL TRIAL: NCT05011929
Title: Comparison of the Effects of Support and Non-support Online Cognitive Behavioural Therapy for Insomnia in Youth: a Randomised Controlled Trial
Brief Title: Comparison of the Effects of Support and Non-support Online CBT-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assisitant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA
Record Dates: First submitted 2021-04-24; First posted 2021-08-18 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A randomised, assessor-blind, parallel group controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online CBT-I with support (individualized feedback and reminders) (Experimental): The mobile-APP based CBT-I consists of 6 weekly session. The treatment is structured and based on the well-established CBT elements for treating insomnia. The treatment components in the CBT-I aim to address the behavioural, cognitive and physiological perpetuating factor of insomnia and include: psycho-education about sleep and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention. reminders and individualized feedback regarding the behavioral strategies will be sent to the participant every week.
  Interventions: Behavioral: Cognitive behavioral therapy
- online CBT-I without support (Active Comparator): same as the experimental arm but without reminders and individualized feedback
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — refer to the arm description

SUMMARY:
Insomnia is the most prevalent sleep problem in children and adolescents and it has been found to predict the development of mental health problems in young adulthood. Cognitive behavioral therapy for insomnia (CBT-I) has been found to be effective in both adults and adolescents. However, limited accessibility and availability of the treatment has only benefited a small proportion of insomnia patients. Therefore, digital CBT-I has been promoted as an alternative way to manage individual's insomnia problems with adequate efficacy. Nonetheless, one of the major limitations of the online self-help intervention is the relatively high drop-out rate and lower compliance compared to the face-to-face modality which the interactive component is less practical in the online intervention. Therefore, the objectives of current study are 1) evaluate the efficacy of mobile-APP based CBT-I in treating youth insomnia, 2) evaluate whether the provision of additional support could further enhance the treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chinese aged 12-24 years old;
* Informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
* Being able to comply with the study protocol;
* Having a DSM-5 diagnosis of insomnia disorder, with a score on Insomnia Severity Index (ISI) >= 9 (suggested cut-off for adolescents)

Exclusion Criteria:

* A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
* Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease);
* Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome;
* Concurrent, regular use of medications(s) known to affect sleep continuity and quality (e.g. hypnotics, steroids);
* In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt);
* Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
* Initiation of or change in antidepressant medication within past 2 months;
* Having been or is currently receiving any structured psychotherapy;
* With hearing or speech deficit;
* Night shift worker.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of insomnia symptoms | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Insomnia Severity Index (ISI) is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change of sleep quality | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of sleep diary measure (total time in bed) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total time in bed (minutes)
Change of sleep diary measure (total sleep time) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (minutes)
Change of sleep diary measure (sleep efficiency) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (%)
Change of sleep diary measure (sleep onset latency) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (minutes)
Change of sleep diary measure (wake after sleep onset) | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (minutes).
Change of daytime sleepiness | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of daytime fatigue | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of quality of life | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of suicidal ideation | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of self-report mood symptoms | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores
Change of dysfunctional beliefs and attitudes about sleep | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of sleep hygiene and practice | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of pre-sleep arousal | Baseline, post-treatment (week 6/at the conclusion of last session) for all participants; and additionally at post-treatment one-month and six-months for those in the two active treatment groups
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No